CLINICAL TRIAL: NCT03650465
Title: Cognitive-behavioral Therapy (CBT) for Generalized Anxiety Disorder: Preliminary Data of Various Contrasting CBT Approaches in a Randomized Clinical Trial
Brief Title: Comparing Different CBT Approaches in GAD
Acronym: CBTforGAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Collaborators: Albert Ellis Institute, New York (Unknown)
Responsible Party: Principal Investigator, Daniel David, Professor, Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BabesBolyaiU
Record Dates: First submitted 2017-12-22; First posted 2018-08-28 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Generalized Anxiety Disorder
Keywords: generalized anxiety; GAD; worry; CBT; REBT; ACT
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CT/BTP (Experimental): Cognitive-behavioral therapy (CBT) in the form of Borkovec's treatment package (CT/BTP for GAD) was derived from Borkovec and Costello's (1993) therapeutic approach, relying on principles of CT for anxiety (A. T. Beck & Emery, 1985) and including applied relaxation. The CT/BTP protocol included several directions as primary goals in therapy: providing a cognitive conceptualization of the problem, identifying and restructuring automatic thoughts, intermediate and core beliefs through cognitive and behavioral techniques (i.e., behavioral experiments), enhancing adaptive behavior (i.e., activity scheduling, dealing with avoidance behavior, social skills training), and using applied relaxation as a coping strategy.
  Interventions: Behavioral: Cognitive-behavioral therapy (CBT)
- REBT (Experimental): Cognitive-behavioral therapy (CBT) in the form of REBT was based on the approach of Dryden & DiGiuseppe (1990), having as a central tenet changing dysfunctional emotions (e.g., anxiety) into functional ones (e.g., healthy anxiety/concern) by changing irrational beliefs into rational beliefs using cognitive, emotive, and behavioral techniques. The structure of an REBT session parallels the CT/BTP session structure including the same elements, but often with a different content. In its elegant/specific form, used here, REBT is focused on changing the core irrational beliefs (i.e., evaluative beliefs/appraisals) seen as the fundamental etiopathogenetic mechanism of GAD.
  Interventions: Behavioral: Cognitive-behavioral therapy (CBT)
- ACT/ABBT (Experimental): Cognitive-behavioral therapy (CBT) in the form of the ACT/ABBT protocol was derived from the principles and techniques proposed by Eifert and Forsyth (2005) and Roemer and Orsillo (2005). From this perspective, GAD is maintained by dysfunctional reactions to internal experiences (i.e., emotions, thoughts, bodily sensations), experiential avoidance, and behavioral restriction, so the treatment aims to address all of these problems. In this sense, ACT/ABBT includes three major treatment goals: (1) education about the nature of anxiety, worry and the role of experiential avoidance; (2) practicing mindfulness and acceptance skills when dealing with disturbing internal experiences; and (3) identifying values and following valued action paths when facing obstacles.
  Interventions: Behavioral: Cognitive-behavioral therapy (CBT)

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy (CBT) — Cognitive-behavioral therapy (CBT)

SUMMARY:
Cognitive-behavior therapy (CBT) is considered the "golden standard" psychotherapy for generalized anxiety disorder (GAD). However, it entails different approaches and blanket statements remain hard to formulate. We conducted a randomized controlled trial to compare the most studied CBT protocol for GAD - Borkovec's treatment package - with two other forms : Rational Emotive Behavior Therapy and Acceptance and Commitment Therapy.

DETAILED DESCRIPTION:
The goal of our present study is to compare the most established and studied CBT protocol for GAD, namely Borkovec's treatment package (BTP) with two other forms of CBT: Rational Emotive Behavior Therapy (REBT; Ellis, 1977) and Acceptance and Commitment Therapy (ACT; Hayes et al., 2012). These two forms of therapy were chosen for both conceptual and practical reasons.

At a conceptual level, we wanted to compare forms of CBT with distinct approaches to dysfunctional thoughts. A fundamental postulate of the cognitive model of psychopathology is that the modification of dysfunctional thoughts (i.e., cognitive change) is central to treating psychological disorders, as "all therapies work by altering dysfunctional cognitions, either directly or indirectly". Both classical Beck's cognitive therapy (CT; Beck, 1976), which is an integrated part in Borkovec's GAD treatment package (CT/BTP), and REBT focus on changing dysfunctional thoughts, but they differ fundamentally in their approach to achieving this change. More specifically, Beck's CT focuses primarily on modifying mental representations of relevant circumstances in the forms of dysfunctional descriptions and inferences (i.e., "cold" cognitions: "I will fail."). REBT on the other hand focuses mainly on "hot" cognitions in the form of evaluations/appraisals (i.e., rational and irrational beliefs), which refer to the ways in which "cold" cognitions/ representations are processed in terms of their relevance for personal well-being (i.e., "I must not fail and it is awful if I fail."). In contrast to both CT and REBT, ACT does not directly attempt to modify the content of the thoughts at all, but aims to change the individual's relationship to dysfunctional beliefs (i.e., the significance of having these beliefs), a process through which cognitions are thought to become "neutralized" (i.e., defused) and the anxiety/distress related to them is reduced or accepted.

At a practical level, we wanted to investigate how different forms of CBT (i.e., REBT and ACT/ABBT) would measure up to the established package based on Borkovec's treatment protocol (CT/BTP).

According to REBT, core irrational beliefs (e.g., "I must not fail and it is awful if I fail."), in interaction to various activating events (e.g., a test situation), generate automatic thoughts in the form of descriptions/inferences (e.g., "I will fail here.") that are then further processed by automatic thoughts in the form of specific irrational beliefs derived from the core irrational beliefs (e.g., "I must not fail here and it is awful if I fail here.") that than further generate anxiety symptoms. In its general form, REBT is focused on changing both core beliefs and automatic thoughts, but in its specific form, used here, REBT is focused on changing the core irrational beliefs seen as the fundamental etiopathogenetic mechanisms of GAD.

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis of generalized anxiety disorder (GAD)

Exclusion Criteria:

* severe major depression
* bipolar disorder
* panic disorder
* substance use/abuse/dependence
* psychotic disorders
* suicidal or homicidal ideation
* organic brain syndrome
* disabling medical conditions
* mental retardation
* concurrent treatment with psychotropic drug
* psychotherapy outside study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-05-16 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Generalized anxiety symptoms | 20 sessions, approximately 16 weeks
  Generalized Anxiety Disorder Questionnaire IV (GAD-Q-IV)
Worry | 20 sessions, approximately 16 weeks
  Penn State Worry Questionnaire (PSWQ)

SECONDARY OUTCOMES:
Automatic thoughts frequency | 20 sessions, approximately 16 weeks
  Automatic Thoughts Questionnaire (ATQ)
Automatic thoughts believability | 20 sessions, approximately 16 weeks
  Automatic Thoughts Questionnaire (ATQ)

CONTACTS AND LOCATIONS:
Locations (1):
- Babes-Bolyai University, Department of Clinical Psychology and Psychotherapy, Cluj-Napoca, Non-US/Non-Canadian, Romania

IPD SHARING:
Plan to Share IPD: Undecided